CLINICAL TRIAL: NCT03690856
Title: DEPREDICT: Clinical and Neurobiological Profile Predictive of Pejorative Outcome of Depression
Brief Title: Clinical and Neurobiological Profile Predictive of Pejorative Outcome of Depression
Acronym: DEPREDICT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 35RC17_8838_DEPREDICT
Record Dates: First submitted 2018-09-18; First posted 2018-10-01 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- depressiv people (Experimental)
  Interventions: Other: inflammatory, neuropsychological and neuroimaging assessment

INTERVENTIONS:
Other: inflammatory, neuropsychological and neuroimaging assessment — Acts add by research:
  pregnancy test; Centralized: IL1, IL6, TNF
  Neuropsychologic tests at M6 and M24:
  Edinburgh Ladder Lateral Test, Direct and Inverse Verbal Empan, Matrices (WAIS IV), Similarities (WAIS IV), Vertebral fluences, STROOP test, TMT test (Delis Kaplan), WCST test, CPT III, WAIS IV (code)

SUMMARY:
Depression is a frequent disease which can be marked by therapeutic resistance. It is described as one of the most disabling disease with high cost for society. World Health Organization pointed out that 350 million people are suffering from depression in the world. This pathology is considered underdiagnosed, with inadequate care resources and stigmatization.

There is a wide range of evidence in current literature that anxiety is one of the most important factors involved in biological mechanism of treatment resistance in depression. To date, there is a lack of knowledge on this topic. A better understanding of the role of anxiety in the maintenance of depressive state will allow to i) identify quickly and more accurately patients at risk of pejorative evolution and ii) develop specific therapeutics targeting this dimension which remain badly controlled with actual therapeutics.

ELIGIBILITY:
Inclusion Criteria:

* Men and women older than 18 years-old;
* Suffering from a Mood Depressive Episode ( according to DSM IV criteria), and-or Mood Depressive recurrent depression (unipolar or bipolar) (<at stage 3 of Thase and Rush). Treatment resistance will be assessed using Thase an Rush Classification and measured with Maudsley Staging Method (Fekadu et al., 2009);
* MADRS score 15;
* Capacity for the patient to receive information on protocol;
* Patient who gave their consent to the protocol.

Exclusion Criteria:

* Contra-indication to MRI
* Patients under social protection or hospitalized without their consent
* Patients suffering from a psychiatric comorbidity such as: schizophrenia, schizo-affective disorder, personality disorder, actual addiction, anorexia-bulimia, obsessive-compulsive disorder;
* Patients suffering from severe intercurrent disease with health prognosis engaged;
* Patients suffering from neurological comorbidity such as: any neurodegenerative disorder (Alzheimer disease, Parkinson disease, Lewy's body disease, multiple sclerosis), any intracranial expansive process.
* Patients with an history of severe cranial injury (with coma);
* Patients with abnormal cerebral MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-11-08 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
MADRS Scale | at 36 months
  Montgomery Äsberg Depression Rating Scale (MADRS): is a scale of depression (diagnosis + follow-up evolution, therapeutic response criteria). It consists of 10 items rated from 0 to 6 from a semi-structured interview, to obtain a total depression score of 0 to 60 (0 no depression, 60 maximum depression intensity). Items evaluate: apparent sadness, expressed sadness, inner tension, reduced sleep, reduced appetite, difficulty concentrating, weariness, inability to feel, pessimistic thoughts, thoughts of suicide ;
STAI YB | at baseline.
  STAI (State Trait Anxiety Inventory) form A and B: is an anxiety scale. The first part concerns state anxiety and consists of a self-questionnaire of 20 items, the subject having to score on a 4-point Likert scale (not at all, little, moderately, much) his current anxiety level. The second part concerns trait anxiety and consists of a self-questionnaire of 20 items, the subject having to score on a 4-point Likert scale (almost never, sometimes, often, almost always) his level of background anxiety. Two scores varying between 10 (minimum anxiety) and 40 (maximum anxiety) are therefore obtained;

SECONDARY OUTCOMES:
MADRS Scale | at 6, 12, 24 months
  Montgomery Äsberg Depression Rating Scale (MADRS): is a scale of depression (diagnosis + follow-up evolution, therapeutic response criteria). It consists of 10 items rated from 0 to 6 from a semi-structured interview, to obtain a total depression score of 0 to 60 (0 no depression, 60 maximum depression intensity). Items evaluate: apparent sadness, expressed sadness, inner tension, reduced sleep, reduced appetite, difficulty concentrating, weariness, inability to feel, pessimistic thoughts, thoughts of suicide ;
MSM | at 6, 12, 24, 36 months
  Maudsley Staging Method (MSM): The Maudsley method allows an evaluation of the degree of pharmacological resistance integrating the main parameters related to the notion of resistance (duration, initial severity of depression, number and types of treatments tested). A treatment must be prescribed at least 6 weeks to be considered as adequate and according to the observed situations an overall score is determined. A score between 3 and 6 characterizes a mild resistance, between 7 and 10, moderate and finally 11 to 15, severe.
AES | at 6, 12, 24, 36 months
  Apathy Assessment Scale (AES) is a scale that evaluates apathy. This is a hetero rating scale from a semi-structured interview by a trained clinician. It has 18 items from 1 (the item is not present) to 4 (the item is very severe). She evaluates cognitive, emotional and behavioral apathy as well as three items of various apathy. The total score ranges from 18 (total absence of apathy) to 72;
ERD | at 6, 12, 24, 36 months
  Depressive Deceleration Scale (DRE): is an instrument that measures the different aspects of idiopathic slowdown related to depression. The specialist evaluates 16 symptoms and scores each of them according to the following rating: 0-normal, 1-doubt on the pathological character of the phenomenon observed, 2-pathological but discrete sign, 3-obvious for any observer, 4-massive;
YMRS | at 6, 12, 24, 36 months
  Young Mania Rating Scale (YMRS): is a scale published in 1978. It is composed of 11 items. It allows to detect and measure the severity of hypomanic episodes in patients with mood disorders. The assessment is based on the patient's condition within 48 hours before the interview and also during the interview. 4 items are rated out of 8 (irritability, speech, idiotic content, aggressive or unstable behavior) and 7 of 4 rated items (mood, motor activity, sleep, interest in sexuality, thinking disorders, presentation, insight );
MADRS | at 6, 12, 24, 36 months
  Montgomery Äsberg Depression Rating Scale (MADRS): is a scale of depression (diagnosis + follow-up evolution, therapeutic response criteria). It consists of 10 items rated from 0 to 6 from a semi-structured interview, to obtain a total depression score of 0 to 60 (0 no depression, 60 maximum depression intensity). Items evaluate: apparent sadness, expressed sadness, inner tension, reduced sleep, reduced appetite, difficulty concentrating, weariness, inability to feel, pessimistic thoughts, thoughts of suicide ;
STAI | at 6, 12, 24, 36 months
  STAI (State Trait Anxiety Inventory) form A and B: is an anxiety scale. The first part concerns state anxiety and consists of a self-questionnaire of 20 items, the subject having to score on a 4-point Likert scale (not at all, little, moderately, much) his current anxiety level. The second part concerns trait anxiety and consists of a self-questionnaire of 20 items, the subject having to score on a 4-point Likert scale (almost never, sometimes, often, almost always) his level of background anxiety. Two scores varying between 10 (minimum anxiety) and 40 (maximum anxiety) are therefore obtained;
Beck | at 6, 12, 24, 36 months
  Short Beck Questionnaire: is a self-assessment scale. The subject is asked to complete the questionnaire by circling the number corresponding to the chosen proposal. It can surround, in a series, several numbers if several propositions are suitable. Each item consists of 4 sentences corresponding to 4 degrees of increasing intensity of a symptom: from 0 to 3. In the stripping, it is necessary to take into account the strongest coast chosen for the same series. The overall score is obtained by adding the scores of the 13 items. The range of the scale is from 0 to 39. The higher the score, the more the subject is depressed.
SHAPS | at 6, 12, 24, 36 months
  SHAPS (Snaith-Hamilton Pleasure Scale, 1995): is a scale that evaluates anhedonia, that is to say the loss of pleasure - among other things in patients with depressive syndrome. This self-questionnaire contains 14 items. The patient is offered 4 types of answers: strongly disagree, disagree, agree, strongly agree. The subjects who complete this ladder are invited to answer based on the ability to experience pleasure in the last days. SHAPS was validated in French in 1997.
HAMA | at 6, 12, 24, 36 months
  HAMA (Hamilton Scale): is a scale of appreciation for anxiety. It has been widely used in clinical trials since 1959. It was translated into French by P. Pichot in 1982. The HAMA includes 14 items covering all areas of psychic anxiety, somatic muscle and visceral disorders cognitive and sleep, depressed mood. Each item is rated from 0 to 4 from the absence to the maximum incapacitating intensity. The overall score ranges from 0 to 60. The evaluator, depending on the items, will take into account the 7 days preceding the interview and the day of the interview included. The contributor is asked to choose the intensity that best suits the patient's clinical condition.
CGI | at 6, 12, 24, 36 months
  CGI (Clinical Global Impression): are three scales that evaluate punctually the severity of the disease, the evaluation of overall improvement and the measurement of the therapeutic index. These three scales were developed as part of the research on schizophrenia and the effect of drugs. These global clinical impressions, however, are not reserved for a specific type of pathology. The first CGI is scored from 0 to 7, 0 corresponding to not evaluated, 1 corresponding to normal, 7 corresponding to among the sickest patients. The second CGI is rated from 0 to 7, 0 corresponding to not evaluated, 1 corresponding to very strongly improved, 7 corresponding to very strongly aggravated. The third CGI for the therapeutic index evaluates the therapeutic effect and the side effects. The CGI are fast (5 minutes).
  The longitudinal clinical evolution will be evaluated by:
  * CGI severity
  * CGI answer
Edinburgh Laterality Test | at 6, 12, 24, 36 months
  Edinburgh Ladder Laterality Test: Assessment of Lateralization. Self-questionnaire with 10 items on the habits of use (right hand or left) for different activities (writing, drawing, throwing, cutting, combing, brushing, cutting, taking a spoon, use of a hammer, screwing ). It allows to calculate a ratio D-G / D + G. According to this ratio, the right or left lateralization is defined;
Empan | at 6, 12, 24, 36 months
  Verbal direct and reverse pitch: measurement of the functioning of the phonological loop (short-term memory) and the central administrator (working memory). The experimenter pronounces series of numbers of increasing size (starting with two-digit series) that the participant must repeat in the same order (for the verbal span location) or in reverse order (for the verbal span) reverse). The examiner notes the maximum size of the correctly recalled series of digits for both types of empan;
Mattis Scale | at 6, 12, 24, 36 months
  Mattis scale: evaluation of cognitive functions. This scale evaluates, from several simple neuropsychological tests, the attention, the initiation, the visuo-constructive capacities, the conceptualization, the temporo-spatial orientation, the mnemic capacities of free recall and recognition. His total score is 144 points. The score is corrected according to age and cultural level;
Verbal fluences | at 6, 12, 24, 36 months
  Verbal fluences: This test tests the action planning abilities, the implementation of semantic memory search strategies and the oral language. The subject has two minutes to give as many words as possible starting with the letter P or in the category of animals. We record the total number of words generated in two minutes in thirty-second increments for each of these conditions.
Stroop Test | at 6, 12, 24, 36 months
  STROOP test: evaluation of executive functions. This test evaluates the resistance to interference, ie the ability of the patient to inhibit some over-learned and automated responses. It consists of three parts: color denomination where the subject must name the color (red, green or blue) of rectangles presented on a board, reading words where the subject must read names of color (red, green or blue) that appear in black characters on a second board and interference where the subject must name the color printed without reading the color name written on a third board. Each board has 100 items. The participant must read column by column. We report for each board the number of correctly named items in 45 seconds. We also calculate an interference index.
Trail Making Test(TMT) Part A and B | at 6, 12, 24, 36 months
  Trail Making Test (TMT) part A and B: evaluation of executive functions. This test assesses mental flexibility and visual exploration capabilities. It is divided into two parts. In Part A, the patient must link the figures in ascending order as quickly as possible. In Part B, the patient must link the numbers and letters in ascending order by following an alternating rule. The time (in seconds) put by the participant to take part A and B and the number of errors will be recorded. For Part B, the examiner also records the number of perseveration errors, that is, when the participant did not follow the alternation rule. Finally, the examiner makes a calculation (time taken for Part A subtracted from the time taken for Part B) to tell whether the participant has a mental flexibility disorder.
  The oral version of this test (Oral Trail Making Test, TMT) will be used for patients over 65 years old with cognitive impairment prior to the depressive episode.
MCST | at 6, 12, 24, 36 months
  Modified Card Sorting test (MCST): assessment of the capacities of conceptualization, attention and mental flexibility. It consists in proposing to the participant a classification of cards according to rules which he must find himself. There are three ranking possibilities that the participant must repeat twice after holding each ranking for six cards. The examiner records the number of correctly found and maintained categories, the total number of errors and the number of perseverative errors.
CPT III | at 6, 12, 24, 36 months
  CPT III (Continuous Performance Test III): assessment of the patient's attentional abilities. This tool is computerized. It is suggested to the patient to hold his attention for 20 minutes. Letters appear on a screen at different speeds and rhythms. The patient must click on the space bar as quickly as possible at each appearance of letters except when the letter X is displayed. The scores evaluate the reaction time as well as the number of errors.
IRM | At baseline and at 36 months
  Neuroimaging

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - CHU angers, Angers
  - CHU de Brest - Hôpital de Bohars, Brest
  - CHU de Nantes - Hotel-Dieu, Nantes
  - CH Henri Laborit, Poitiers
  - CH Guillaume Regnier, Rennes
  - EPSM du Morbihan, Saint-Avé
  - CH Saint-Malo, St-Malo
  - CHU de Tours, Clinique Psychiatrique Universitaire, Tours